CLINICAL TRIAL: NCT00416546
Title: A Double Blind, Randomized, Placebo-Controlled Study of AEB071 in Healthy Volunteers to Evaluate the Safety/Tolerability of 14 Day Multiple-Dose AEB071 and Measure the Effect of Ethnicity on Pharmacokinetics, Pharmacodynamics and Safety/Tolerability in Caucasian and Japanese Subjects Receiving Single and Multiple Doses of AEB071
Brief Title: Safety of AEB071 in Healthy Volunteers and to Compare the Ethnicity, Metabolic, and Safety Effects Between Caucasian and Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAEB071A2113
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: Healthy Caucasians; Healthy Japanese subjects; Immunosuppressant; early T-cell activation blockers; inhibition of protein kinase C
MeSH Terms: interventions — sotrastaurin

INTERVENTIONS:
Drug: AEB071

SUMMARY:
This is a study to assess the safety effects after multiple doses of AEB071 in healthy volunteers and to compare the ethnicity, metabolic, and safety effects between Caucasian and Japanese healthy subjects receiving single and multiple doses of AEB071.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects having provided written, informed, consent before entering the study. Light smokers (≤10 cigarettes/day) will be eligible for inclusion in this study. Smokers will be defined as any subject who reports cigarette use or has a urine cotinine greater than 500 ng/mL.
* Female subjects must be either surgically sterilized at least 6 months or practicing an acceptable form of birth control (i.e. double barrier method - intrauterine device plus condom, spermicidal gel plus condom).
* Subjects must have a body weight between 45 and 90 kg and a body mass index (BMI) between 18-28 kg/m2.
* Japanese subjects of 1st, 2nd, or 3rd generation ethnic origin or Caucasian.
* Japanese subjects will be defined as being of Japanese ethnicity with all 4 grandparents of Japanese descent. Generations will be defined as follows:

  * 'First generation' Japanese are subjects who were born in Japan to parents of Japanese ethnicity.
  * 'Second generation' will be defined as subjects who were born outside of Japan to 1st generation Japanese parents.
  * 'Third generation' will be defined as subjects born outside of Japan to 2nd generation Japanese parents, i.e. 4 grandparents from Japan but both parents and subject born elsewhere.
* Caucasians are defined as subjects with all four grandparents of European descent.

Exclusion Criteria:

* Presence and/or history of a clinically significant illness within two weeks prior to dosing, history of drug or alcohol abuse within the 12 months prior to dosing, use of any prescription drug or over-the-counter (OTC) medication (acetaminophen is acceptable) within 14 days prior to dosing.
* Presence of a clinically significant systemic illness, active infectious process (viral or bacterial), e.g., cold sore, or documented drug allergies that may deteriorate or affect the subject's safety or ability to cooperate during the study.
* Laboratory or clinical evidence suggestive of liver or renal disease, history of heart disease, history of autonomic dysfunction (e.g. history of fainting, orthostatic hypotension, sinus arrhythmia), history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated), history of major gastrointestinal disease, history or clinical evidence of pancreatic injury or pancreatitis
* Subjects with a resting heart rate < 50 beats per minute (bpm)
* Subjects with systolic blood pressure < 90 or diastolic blood pressure < 50.
* Subjects with lymphocyte counts less than 1200/mm3 or total white blood cell (WBC) greater than 10000/mm3 at baseline
* A past medical history of clinically significant electrocardiogram (ECG) abnormalities or a family history of a prolonged QT-interval syndrome.
* Subjects who intend to or have received any live attenuated vaccines 4 weeks prior to or during the study period.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2006-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacokinetics between healthy Caucasian and Japanese subjects after a single oral dose of AEB071
To compare the pharmacokinetics between healthy Caucasian and Japanese subjects after 7 days of oral, daily doses of AEB071
To compare the safety and tolerability of single and multiple oral doses of AEB071 in healthy Japanese and Caucasian subjects

SECONDARY OUTCOMES:
To compare the dose response, temporal course and effect of AEB071 on lymphocyte proliferation after single oral doses of AEB071 in healthy Caucasian and Japanese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis
Locations (1):
- Novartis Investigative Site, Dorval, Quebec, Canada